CLINICAL TRIAL: NCT01056718
Title: Effects of Nebivolol on Exercise Tolerance and Left Ventricular Systolic and Diastolic Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Research (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, James Stokes, MD, Cardiologist Mercy Hospital, Mercy Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BYS-MD-32
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Hypertension
Keywords: Diastolic Function; Nebivolol
MeSH Terms: conditions — Hypertension | interventions — Nebivolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nebivolol treatment (Other): 10 week open label nebivolol treatment.
  Interventions: Drug: Nebivolol

INTERVENTIONS:
Drug: Nebivolol — Initial dose of 5 mg titrated (doubling of previous dose) to optimal blood pressure. The dose was titrated by doubling the previous dosage to achieve BP less than or equal to 130/80 mm Hg at 2 weeks and 4 weeks. The mean dose of nebivolol used week 4 through week 10 was 7.8 mg. It should be noted that nebivolol was added to the subject's existing stable antihypertensive regimen which included a mean of 2 other medications.

SUMMARY:
The goal of this pilot study is to effectively treat hypertension in subjects with either known or newly diagnosed hypertension and concurrent evidence of diastolic dysfunction. Due to the unique properties of nebivolol, it is hypothesized that there will be improvements in left ventricular (LV) systolic and diastolic function manifesting as increase exercise capacity in this patient population with primarily LV diastolic dysfunction. The present study was performed to determine the effects of nebivolol on blood pressure, exercise tolerance and parameters of left ventricular systolic and diastolic function in a group of hypertensive patients with echocardiographic evidence diastolic dysfunction.

DETAILED DESCRIPTION:
Prior to the initiation of Nebivolol and after 10 weeks of Nebivolol therapy, subjects underwent a resting 2D echocardiogram including routine sampling of mitral valve (MV) inflow and LV tissue Doppler imaging as well as a symptom limited exercise treadmill stress test with echocardiographic imaging. Primary endpoints were 1) changes in systolic blood pressure before and after 10 weeks of treatment and 2) changes in exercise capacity as determined by exercise duration and metabolic equivalent (MET) level before and after treatment. Secondary endpoints were changes in exercise hemodynamics and Doppler echocardiographic parameters of LV systolic and diastolic function and quality of life before and after 10 weeks of nebivolol treatment. Subjects completed an EuroQol (EQ-SD) Quality of Life questionnaire which is a standardized measure of health status developed by the EuroQol group as a simple general measure of health at baseline and at conclusion of the 10 week trial period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis (new or established) hypertension, defined by serial measurements >/= 140/90
* Evidence of diastolic dysfunction on echocardiography measured by tissue Doppler

Exclusion Criteria:

* Severe bronchospastic disease/ reactive airway disease
* Inability to tolerate beta blocker therapy including: >1st degree atrioventricular (AV) block, symptomatic hypotension, symptomatic bradycardia,
* Subjects with physical limitations that would prevent them from participating in an exercise treadmill test
* Age <18 or >90 years
* Those with life expectancy <1 year
* Subjects with class III/IV New York Heart Association (NYHA) heart failure symptoms
* Chronic Kidney Disease 3 or greater (CrCl <30 cc/min)
* Subjects with active ischemia or evidence of ischemia on initial stress echocardiography

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-11; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A. Stokes, M.D., Principal Investigator — St. John's Mercy Heart & Vascular
Locations (1):
- St. John's Mercy Cardiovascular Research, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from the outpatient office at Mercy St. Louis between January 2010 and August 2012. The inclusion criteria were new or established hypertension as defined by serial BP measurements greater than or equal to 140/90 and evidence of left ventricular (LV) diastolic dysfunction as defined by a routine Doppler within a year of enrollment.
Period: Overall Study
Arm/Group | Nebivolol Treatment
Started | 53
Completed | 50
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Ischemia on baseline stress test | 1

BASELINE CHARACTERISTICS:
Groups:
- Nebivolol Treatment: All subjects will begin an initial dosage of 5mg of Nebivolol titrated (doubling of previous dose) to optimal blood pressure below 130/80 at 2 and 4 weeks after treatment initiation.
  Nebivolol: Initial dose of 5 mg titrated (doubling of previous dose) to optimal blood pressure.
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 53
BMI [Mean (Standard Deviation); unit: kg/m2] | 31 (5)
Resting Systolic BP [Mean (Standard Deviation); unit: mm Hg] | 145 (19)
Exercise Duration [Mean (Standard Deviation); unit: seconds] | 385 (174)
Metabolic Equivalent [Mean (Standard Deviation); unit: Mets] — One MET is defined as 3.5 mL 02 uptake/kg per minute
  Mets | 6.2 (3.1)
Resting Diastolic BP [Mean (Standard Deviation); unit: mm Hg] | 79 (11)
Peak Stress Systolic BP [Mean (Standard Deviation); unit: mm Hg] | 178 (23)
Peak Stress Diastolic BP [Mean (Standard Deviation); unit: mm Hg] | 75 (15)
Resting Heart Rate [Mean (Standard Deviation); unit: Beats per Minute] | 69 (11)
Stress Heart Rate [Mean (Standard Deviation); unit: Beats per Minute] | 136 (24)
Resting Ejection Fraction (EF) [Mean (Standard Deviation); unit: Percent of LV end diastolic volume] — Ejection fraction = LV end diastolic volume - LV end systolic volume divided by LV end diastolic volume X 100
  Percent of LV end diastolic volume | 61 (10)
Stress EF [Mean (Standard Deviation); unit: Percent of LV end diastolic volume] | 67 (10)
Resting Stroke Volume [Mean (Standard Deviation); unit: ml] | 46 (15)
Stress Stroke Volume [Mean (Standard Deviation); unit: ml] | 47 (13)
Resting Cardiac Output [Mean (Standard Deviation); unit: L per minute] | 3.1 (1.1)
Stress Cardiac Output [Mean (Standard Deviation); unit: L per minute] | 5.6 (2.2)
LV End Diastolic Diameter [Mean (Standard Deviation); unit: cm] | 4.7 (0.5)
LV End Systolic Diameter [Mean (Standard Deviation); unit: cm] | 3.0 (0.8)
LV Mass [Mean (Standard Deviation); unit: grams] | 163 (52)
Mitral Valve Inflow (E) Velocity [Mean (Standard Deviation); unit: cm/s] | 77 (24)
Mitral Valve Inflow (A) Velocity [Mean (Standard Deviation); unit: cm/s] | 91 (21)
Mitral Valve E/A Ratio [Mean (Standard Deviation); unit: Ratio] — Mitral valve doppler E velocity to A velocity
  Ratio | .86 (.18)
Mitral Valve Deceleration Time [Mean (Standard Deviation); unit: ms] | 229 (62)
Mitral Valve Tissue Doppler Velocity (e') [Mean (Standard Deviation); unit: cm/s] | 7.6 (1.9)
Mitral Valve Tissue Doppler Velocity (a') [Mean (Standard Deviation); unit: cm/s] | 11.8 (2.9)
E/e' Ratio [Mean (Standard Deviation); unit: Ratio] — Mitral Valve E velocity to tissue doppler e' velocity
  Ratio | 10.8 (4.7)
Pulmonary Vein Peak Systolic Velocity [Mean (Standard Deviation); unit: cm/s] | 62 (13)
Pulmonary Vein Peak Diastolic Velocity [Mean (Standard Deviation); unit: cm/s] | 47 (13)
Quality of Life [Mean (Standard Deviation); unit: units on a scale] — Subjects completed an EuroQol (EQ-SD) Quality of Life questionnaire which is a standardized measure of health status developed by the EuroQol group as a simple general measure of health. The EuroQol, records the subject's self reported assessment of his/her overall health on a vertical, visual analogue scale where 100 is "the best imaginable health state" and 0 is the "worst imaginable health state".
  units on a scale | 77 (12)

OUTCOME MEASURES:

1. Primary Outcome: Resting Systolic BP
Time Frame: 10 Weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
mm Hg | 135 (17)
Statistical Analysis 1: Comparison: Nebivolol Treatment; Nebivolol treatment group refers to 50 patients that completed 10 weeks of open label nebivolol treatment. Results were compared using paired T-tests in a pre - post study design before and after 10 weeks of treatment. Each subject served as his/her own control; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Primary Outcome: Exercise Duration
Time Frame: 10 Weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
Seconds | 419 (180)
Statistical Analysis 1: Comparison: Nebivolol Treatment; Nebivolol treatment group refers to 50 patients that completed 10 weeks of open label nebivolol treatment. Results were compared using paired T-tests in a pre - post study design before and after 10 weeks of his/her treatment. Each subject served as own control; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

3. Primary Outcome: Metabolic Equivalent (METS) Level
Description: METs is a measure of exercise capacity. One MET is defined as 3.5 mL 02 uptake/kg per minute which is the resting oxygen uptake in a sitting position. The Bruce protocol consisted of successive 3 minute stages each of which requires the subject to walk at a faster speed and higher grade of incline. Each stage is assigned a MET level. The achieved exercise capacity in METs has been shown to be predictive in older adult population of survival with higher MET levels associated with improved survival.
Time Frame: 10 Weeks
Measure: Mean (Standard Deviation); unit: METS
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
METS | 6.7 (3.2)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

4. Secondary Outcome: Diastolic BP
Time Frame: 10 Week
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
mm Hg | 76 (9)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .078, t-test, 2 sided

5. Secondary Outcome: Peak Stress Systolic BP
Time Frame: 10 Week
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
mm Hg | 171 (26)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .186, t-test, 2 sided

6. Secondary Outcome: Peak Stress Diastolic BP
Time Frame: 10 Week
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
mm Hg | 68 (17)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

7. Secondary Outcome: Resting Heart Rate
Time Frame: 10 Week
Measure: Mean (Standard Deviation); unit: Beats per Minute
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
Beats per Minute | 65 (9)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

8. Secondary Outcome: Stress Heart Rate
Time Frame: 10 Week
Measure: Mean (Standard Deviation); unit: Beats per Minute
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
Beats per Minute | 118 (24)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.06, t-test, 2 sided

9. Secondary Outcome: Resting EF
Time Frame: 10 Weeks
Measure: Mean (Standard Deviation); unit: Percent of LV end diastolic volume
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
Percent of LV end diastolic volume | 63 (9)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

10. Secondary Outcome: Stress EF
Time Frame: 10 Week
Measure: Mean (Standard Deviation); unit: Percent of LV end diastolic volume
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
Percent of LV end diastolic volume | 72 (10)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

11. Secondary Outcome: Resting Stroke Volume
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
ml | 48 (14)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.85, t-test, 2 sided

12. Secondary Outcome: Stress Stroke Volume
Time Frame: 10 week
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
ml | 51 (16)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.40, t-test, 2 sided

13. Secondary Outcome: Resting Cardiac Output
Time Frame: 10 week
Measure: Mean (Standard Deviation); unit: L per minute
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
L per minute | 3.0 (0.9)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.64, t-test, 2 sided

14. Secondary Outcome: Stress Cardiac Output
Time Frame: 10 week
Measure: Mean (Standard Deviation); unit: L per minute
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
L per minute | 5.3 (1.7)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.49, t-test, 2 sided

15. Secondary Outcome: LV End Diastolic Diameter
Time Frame: 10 week
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
cm | 4.8 (0.6)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.47, t-test, 2 sided

16. Secondary Outcome: LV End Systolic Diameter
Time Frame: 10 week
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
cm | 3.1 (0.7)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.55, t-test, 2 sided

17. Secondary Outcome: LV Mass
Time Frame: 10 week
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
grams | 167 (47)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.64, t-test, 2 sided

18. Secondary Outcome: Mitral Valve Inflow (E) Velocity
Time Frame: 10 Week
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
cm/s | 85 (21)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

19. Secondary Outcome: Mitral Valve Inflow (A) Velocity
Time Frame: 10 Week
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
cm/s | 90 (23)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .526, t-test, 2 sided

20. Secondary Outcome: Mitral Valve E/A Ratio
Description: mitral valve doppler E velocity to A velocity
Time Frame: 10 Week
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
Ratio | 0.97 (0.31)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

21. Secondary Outcome: Mitral Valve Deceleration Time
Time Frame: 10 Week
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
ms | 227 (55)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .925, t-test, 2 sided

22. Secondary Outcome: Mitral Valve Tissue Doppler Velocity (e')
Time Frame: 10 Week
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
cm/s | 8.7 (2.6)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

23. Secondary Outcome: Mitral Valve Tissue Doppler Velocity (a')
Time Frame: 10 Week
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
cm/s | 11.5 (2.9)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .458, t-test, 2 sided

24. Secondary Outcome: E/e' Ratio
Time Frame: 10 Week
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
Ratio | 10.5 (4.4)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .561, t-test, 2 sided

25. Secondary Outcome: Pulmonary Vein Peak Systolic Velocity
Time Frame: 10 Week
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
cm/s | 63 (10)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .734, t-test, 2 sided

26. Secondary Outcome: Pulmonary Vein Peak Diastolic Velocity
Time Frame: 10 Week
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
cm/s | 51 (16)
Statistical Analysis 1: Comparison: Nebivolol Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .129, t-test, 2 sided

27. Secondary Outcome: Quality of Life
Description: Quality of life was assessed by a visual analogue scale before and after 10 weeks of nebivolol. The subjects self reported assessment of his/her overall health was recorded on a vertical visual analogue scale where 100 is the "best imaginable health state" and 0 is the "worst imaginable health state".
Time Frame: 10 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nebivolol Treatment
Number analyzed (Participants) | 50
units on a scale | 78 (15)

ADVERSE EVENTS:
Time Frame: Patients were monitored for 10 weeks for any adverse side effects resulting in discontinuation or decrease in nebivolol dosage after the titration period. They were also monitored for cardiovascular events during the treatment period.
Groups:
- Starting on 5 mg of Nebivolol Then Titrated: all subjects will begin an initial dosage of 5mg of Nebivolol titrated (doubling of previous dose) to optimal blood pressure below 130/80 at 2 and 4 weeks after treatment initiation.
  Nebivolol: Initial dose of 5 mg titrated (doubling of previous dose) to optimal blood pressure.
Arm/Group | Starting on 5 mg of Nebivolol Then Titrated
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

LIMITATIONS AND CAVEATS:
There was no placebo control. All patients received nebivolol and served as their own control before and after treatment. This study had a small study population and short duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No